CLINICAL TRIAL: NCT01269814
Title: The Impact of Rockall Risk Scoring System on Timing of Endoscopy, Length of Hospital Stay, Morbidity and Mortality in Patients With Upper Gastrointestinal System Bleeding
Brief Title: The Impact of Rockall Risk Scoring System on Management of Upper Gastrointestinal System Bleeding
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Bakirkoy Dr. Sadi Konuk Research and Training Hospital (Other Government)
Responsible Party: Principal Investigator, Murat Gonenc, Medical Doctor, Bakirkoy Dr. Sadi Konuk Research and Training Hospital
Other Study IDs: Rockall-GIH
Record Dates: First submitted 2010-12-30; First posted 2011-01-04 (Estimated); Last update posted 2012-10-17 (Estimated); Status verified 2012-10

CONDITIONS: Gastrointestinal Hemorrhage
Keywords: Gastrointestinal bleeding; Emergency endoscopy; Rockall Risk Scoring System
MeSH Terms: conditions — Gastrointestinal Hemorrhage | interventions — Gastroscopy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Go-home group: The patients with a Rockall score of 0 or 1 will be prescribed medical therapy, and will be scheduled for elective gastroscopy.
  Interventions: Procedure: Gastroscopy

INTERVENTIONS:
Procedure: Gastroscopy — Gastroscopy

SUMMARY:
The patients who admit to emergency department with upper gastrointestinal system bleeding will undergo a clinical evaluation with Rockall Risk Scoring System. The patients with Rockall score of 1 or less will be discharged with medical treatment, and will have an elective upper gastrointestinal endoscopy in the end of the 30th day. The impact of Rockall Risk Scoring System on assessing the necessity of emergency endoscopy, length of hospital stay, morbidity, and mortality in low-risk patients will be evaluated.

DETAILED DESCRIPTION:
The patients who admit to emergency department with symptoms of upper gastrointestinal system bleeding will undergo a clinical evaluation. First, diagnosis of upper gastrointestinal system bleeding will be established by combined physical examination and nasogastric tube application. After a certain diagnosis, all of the patients will be scored according to Rockall Risk Scoring System. The patients with a 1 or less Rockall score will have conservative treatment including mucosal protective agent (sucralfat), proton pump inhibitors (omeprazole, lansoprazole, pantoprazole), and hemodynamic monitorization. Should Rockall score and hemodynamic parameters remain unchanged or get improved in the end of 6 hours after admission, oral feeding will be started and the patient will be discharged with anti-ulcer medication (mucosal protective agent and proton pump inhibitor, PO). These patients will be scheduled for upper gastrointestinal endoscopy at 30th day. The patients who have: an initial Rockall score of 2 or greater, an increase in Rockall score or deterioration in hemodynamic parameters during observation, will have emergency endoscopy and will be excluded from the study.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of upper gastrointestinal system bleeding
* Rockall score of 1 or less
* Volunteers
* Agreement with the terms of informed consent

Exclusion Criteria:

* Uncertain clinical diagnosis of upper gastrointestinal system bleeding
* Rockall score of 2 or greater
* Deterioration in hemodynamic parameters during follow-up
* Unwilling patients to join the study
* Disagreement with the terms of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients older than 18 years with upper gastrointestinal hemorrhage.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2010-12; Primary Completion 2012-12 (Estimated); Study Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
The necessity of emergency endoscopy. | 1 month

SECONDARY OUTCOMES:
Morbidity | 1 month
Mortality | 1 month
Length of hospital stay | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Halil Alis, MD, Study Director — Dr. Sadi Konuk Training and Research Hospital
Locations (1):
- Dr. Sadi Konuk Training and Research Hospital, Istanbul, Turkey (Türkiye)